CLINICAL TRIAL: NCT05249062
Title: A Non-randomised Pilot Study of the Smart and Healthy Ageing Through People Engaging in Supportive Systems (SHAPES) Digital App and Platform for Supporting Medicines Optimisation in Older Individuals With Multiple Long-term Conditions
Brief Title: SHAPES: Supporting Multimorbid Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Michael Scott (Other Government)
Collaborators: Mid and East Antrim Agewell Partnership (MEAAP) (Unknown); University of Nicosia (Other); Vicomtech (Unknown); TREE Technology S.A. (Unknown); National University of Ireland, Maynooth (Other); Gnomon Informatics S.A. (Unknown); Edgeneering LDA (Unknown); Fraunhofer-Institute of Toxicology and Experimental Medicine (Other); University of Ulster (Other)
Responsible Party: Sponsor-Investigator, Prof Michael Scott, Prof Michael Scott, Northern Health and Social Care Trust
Organization: Northern Health and Social Care Trust (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NT21-SHAPES; 857159 (Other Grant/Funding Number: European Union's Horizon 2020 research&innovation programme); 284743 (Other: IRAS number)
Record Dates: First submitted 2021-12-15; First posted 2022-02-21 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): The intervention being piloted in this study is a novel system of supporting older individuals with multiple long-term conditions to self-manage their chronic conditions through the daily use of a digital health product that can also facilitate the remote monitoring of a person's health status.
  Interventions: Device: SHAPES app

INTERVENTIONS:
Device: SHAPES app — Participants will be asked to use the app and connected devices daily for 3 months.

SUMMARY:
The Smart & Healthy Ageing through People Engaging in Supportive Systems (SHAPES) Innovation Action is a Horizon 2020, EU-wide project looking at how technology can enable the older population to live healthier lives at home. It involves the development, piloting and deployment of a large scale, EU-standardised open platform. This platform will integrate with a wide-range of technological, organisational, clinical, educational and societal solutions seeking to facilitate long-term healthy and active aging.

Within this project are 7 pilot themes investigating various potential uses of the platform, in Northern Ireland we are leading on medicines control and optimisation.

This pilot is focused on identifying, managing and improving deficiencies in adherence to medicines and treatments of older individuals living with permanent or temporary reduced functions or capabilities due to chronic, age-related illnesses and living at home. Digital Solutions (including blood pressure monitors, pulse oximeters, weight scales and glucometers) will be used to enable self-monitoring of the individual's physiological parameters. Data will also be used to develop an algorithm to help predict decompensations in participants with heart failure and dynamic personal ranges will also be developed. In the future this may enable early opportunities to adjust medicines and treatments so as to deliver safer and more effective use of medicines in-home, however, in this pilot there will be no changes to treatment.

The target population is composed of older individuals (+65 years) living at home with heart failure and/or diabetes. We aim to recruit 30 people (for 3 months) to our pilot in Northern Ireland. We are working closely with colleagues in Spain, Czech Republic, Cyprus and Germany to run similar pilots within their healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Northern Health and Social Care Trust service user
* ≥60 years
* Diagnosed with heart failure and/or diabetes mellitus (treatment includes regular self-monitoring of blood glucose)
* Lives at home or in supported living accommodation (category 1 or 2).

  * Category 1 - self-contained accommodation for the more active elderly, which may include an element of scheme supervisor support and/or additional communal facilities
  * Category 2 - scheme supervisor supported self-contained accommodation for the less active elderly, which includes the full range of communal facilities
* Has stable self-reported Wi-Fi connection at home
* Has access to an appropriate android smartphone or tablet
* Android device running version 8 or above; supports Wi-Fi; supports BLE; front facing camera for facial recognition
* Self-reported stable disease state, the participant feels well enough to take part in the pilot
* Self-reported confident user of smartphone/tablet

Exclusion Criteria:

* Participant report of cognitive impairment
* Wears an electronic medical device or implant (e.g. pacemaker, electrocardiogram)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Participants' engagement with the SHAPES app during the pilot | 3 months (end of pilot)
  The number of times the app is opened per day

SECONDARY OUTCOMES:
Participants' user experience with the SHAPES app | 3 months (end of pilot)
  Measured using the User Experience Questionnaire -short version (UEQ-S) A score of -3 to 3 is generated for each participant. A higher score indicates a positive user experience.
Usability of the SHAPES app | 3 months (end of pilot)
  Measured using the System Usability Scale A score of 0 to 100 is generated for each participant. A higher score indicates better usability.
Number and rate of successful registrations of each clinical parameter per participant, per day | 3 months (end of pilot)
  Measured by determining the number of successful registrations of each clinical parameter, per participant, per day (i.e., actual measure of clinical parameter is not relevant to this outcome).
  Findings presented as a percentage of total number of expected registrations a day i.e., 0 to 100% success rate for each parameter.
Number and rate of control limits (upper and lower) successfully generated by the 'Vitals Control' analytic tool per person | 3 months (end of pilot)
  Rate defined as number of pairs of limits generated per week during the pilot
Number and rate of heart failure decompensation prediction (HFPred) risk scores successfully generated per person | 3 months (end of pilot)
  Rate defined as number of scores generated per week during the pilot
Change in hospitalisation rate per person (hospitalisations/month) and A&E attendance rate (attendance/month) | Three months prior to baseline compared with 3 months during the pilot
  Change in hospitalisation rate per person (hospitalisations/month) and A&E attendance rate (attendance/month)
Participants' self-reported medication adherence | Baseline and 3 months (end of pilot)
  Measured using the Medication Adherence Report Scale (MARS) A score between 5 and 25 is generated for each participant. A higher score indicates better adherence.
Participants' beliefs about medicines | Baseline and 3 months (end of pilot)
  Measured using the Belief's about Medicines Questionnaire (BMQ) There are two scales in this outcome. The Necessity Scale assesses beliefs about personal need for medicines. The Concerns Scale assesses medication concerns.
  A score between 5-25 is generated for each scale for each participant.
  The two scores are amalgamated to produce the Necessity Concerns Differential (subtract Concerns Score from the Necessity Score) to give a score between -20 and 20. Higher scores indicate stronger beliefs in the necessity of medication and fewer concerns about taking it.
Correlation between participants' self-reported medication adherence and beliefs about medicines | 3 months (end of pilot)
  The correlation between participants' self-reported medication adherence as measured using the Medication Adherence Report Scale (see outcome 8) and their Belief's about Medicine's Questionnaire- Necessity Concerns Differential (see outcome 9) will be measured statistically using an appropriate correlation coefficient (Pearson correlation coefficient OR Spearman's Rank Order correlation coefficient).
  Note: the study will not be powered to show statistical significance of the correlation but will indicate a possible strength and direction of the relationship.
Number and rate (score/week) of heart failure decompensation prediction (HFPred) risk scores successfully generated per person during the pilot | 3 months (end of pilot)
  Number and rate of heart failure decompensation scores generated
Correlation between HFPred scores and unscheduled care during the pilot | 3 months (end of pilot)
  An appropriate statistical test will be performed to determine whether, or not, there is a correlation between incidence of unscheduled care use (unscheduled care defined as composite of hospitalisations, A&E attendances, specialist contacts, out-of-hours contacts) and heart failure decompensation prediction (HFPred) risk scores.
  Note: the study will not be powered to show statistical significance of the correlation but will indicate a possible strength and direction of the relationship.
Health-related quality of life as measured using the EuroQol 5 dimension 5 level (EQ-5D-5L) descriptive system and visual analogue scale | Baseline and 3 months (end of pilot)
  The EuroQol 5 dimension 5 level (EQ-5D-5L) questionnaire will be used to describe the five dimensions of health related quality of life (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION) for each participant.
  Each of the five dimensions comprising the EQ-5D descriptive system is divided into five levels of perceived problems:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems.
  A unique health state is defined by combining one level from each of the five dimensions. A total of 3125 possible health states is defined in this way. Each state is referred to by a 5-digit code.
  The visual analogue scale records the participants' self-rated health on a vertical visual analogue scale between 0 and 100. Higher scores indicate better perceived health.
Exploration of healthcare practitioners' views on integration and alignment of the SHAPES platform and Digital Solutions with current care pathways | 3 months (end of pilot)
  Measured via qualitative interview
Exploration of healthcare practitioners' views about their trust and acceptance of the SHAPES platform and Digital Solutions | 3 months (end of pilot)
  Measured via qualitative interview
Exploration of participants' views about their trust and acceptance of the SHAPES app | 3 months (end of pilot)
  Measured via qualitative interview
Exploration of user engagement behaviors | 3 months (end of pilot)
  Measured via cross-comparative exploratory analysis of user event logs and qualitative interviews with participants.

OTHER OUTCOMES:
Participants' self-efficacy as measured using the General Self-Efficacy Scale | Baseline, 3 months (end of pilot) and follow-up (further 3 months)
  Measured using the general self-efficacy scale. A score between 10 and 40 is generated, with a higher score indicating more/better self-efficacy.
Participants' extent of social support | Baseline, 3 months (end of pilot) and follow-up (further 3 months)
  Measured using the Oslo Social Support Scale (OSSS-3). A score between 3 and 14 is generated with high values representing strong levels and low values representing poor levels of social support.
Participants' health literacy | Baseline, 3 months (end of pilot) and follow-up (further 3 months)
  Measured using the Single-item Health Literacy Measure (HLM1)
Participation in society | Baseline, 3 months (end of pilot) and follow-up (further 3 months)
  Measured using non-validated participation questions
Participants' quality of life score as measured using the World Health Organization Brief Quality of life tool (WHOQOL-BREF) | Baseline, 3 months (end of pilot) and follow-up (further 3 months)
  Measured using the WHOQOL-BREF. A score between 0 and 100 is generated. Higher score indicates a better quality of life.
Health-related quality of life as measured using the EuroQol 5 dimension 5 level (EQ-5D-5L) descriptive system and visual analogue scale | Baseline and 3 months (end of pilot)
  The EuroQol 5 dimension 5 level (EQ-5D-5L) questionnaire will be used to describe the five dimensions of health related quality of life (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION) for each participant.
  Each of the five dimensions comprising the EQ-5D descriptive system is divided into five levels of perceived problems:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems.
  A unique health state is defined by combining one level from each of the five dimensions. A total of 3125 possible health states is defined in this way. Each state is referred to by a 5-digit code.
  The visual analogue scale records the participants' self-rated health on a vertical visual analogue scale between 0 and 100. Higher scores indicate better perceived health.
Usability of the SHAPES app | 3 months (end of pilot)
  Measured using the System Usability Scale A score of 0 to 100 is generated for each participant. A higher score indicates better usability.
Technology Acceptance | 3 months (end of pilot)
  Measured using technology acceptance questions
Exploration of participants' views about their trust and acceptance of the SHAPES platform and Digital Solutions | 3 months (end of pilot)
  Measured via qualitative interview
Exploration of healthcare practitioners' views about their trust and acceptance of the SHAPES platform and Digital Solutions | 3 months (end of pilot)
  Measured via qualitative interview
Change in health service utilisation for unscheduled care related to heart failure and diabetes | 3 months prior to baseline and 3 months (end of pilot)
  Measured by number of: hospitalisations; A&E attendances; out of hours contacts; contacts with specialist services.
  * Number of hospitalisations
  * A&E attendances
  * Out of hours contacts
  * Contacts with specialist services
Economic impact of the intervention | 3 months (end of pilot)
  as measured by comparing the cost of the intervention (devices, SHAPES platform and digital solutions; staffing) versus the cost of unscheduled care related to heart failure and diabetes during the pilot.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scott, Principal Investigator — Northern Health and Social Care Trust
Locations (1):
- Medicines Optimisation Innovation Centre, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT05249062/Prot_003.pdf